CLINICAL TRIAL: NCT06911736
Title: Effect of the Postoperative Trendelenburg Position on Chronic Subdural Hematoma Recurrence: a Clinical Trial
Brief Title: Effect of the Postoperative Trendelenburg Position on Chronic Subdural Hematoma Recurrence
Acronym: POTHeR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Ignacio Alberto Gonzalez Borrero, Neurosurgeon, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102024
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-05

CONDITIONS: Chronic Subdural Hematoma; Trendelenburg; Recurrence; Mortality; Prognosis; Clinical Trials
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The nature of this intervention did not allow for masking of treatment allocation, so both patients and their care team knew their assigned arm, while outcome assessors and data analysts remained blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control group received the usual postoperative care for patients with CSH, which consisted of strict neurological monitoring for at least 24 hours in an inpatient ward or a more complex setting depending on the patient's clinical condition. The head of the patient was positioned neutral (0°), as were the lower limbs, according to institutional care guidelines. The drain (a latex-gloved reservoir or Hemovac drain) was positioned inferior to the head to promote drainage of any subdural debris. Negative pressure was not used except in patients with Hemovac and a subgaleal drain. Typically, after 24 hours of clinical monitoring and symptom improvement, the drain was removed, and the patient was sent home with recommendations and warning signs, if the patient's clinical condition permitted. Postoperative follow-up imaging was not routinely performed as there was no evidence of clinical benefit.
- Trendelenburg (Experimental): In addition to the management described above, the postoperative position was modified in the intervention group (trendelenburg). After admission to the hospital unit (general ward, special care, or intensive care unit), the patient's position was adjusted with a 30° leg elevation and a 10° downward head tilt. Proper positioning was verified with a goniometer. This position was maintained until the drains were removed, and the patient was then positioned according to usual care. If the patient decided to get out of bed, the nurse occluded the drains and reopened them when the patient returned to the position described for each group.
  Interventions: Other: Trendelenburg position

INTERVENTIONS:
Other: Trendelenburg position — In addition to the management described above, the postoperative position was modified in the intervention group (trendelenburg). After admission to the hospital unit (general ward, special care, or intensive care unit), the patient's position was adjusted with a 30° leg elevation and a 10° downward head tilt. Proper positioning was verified with a goniometer. This position was maintained until the drains were removed, and the patient was then positioned according to usual care. If the patient decided to get out of bed, the nurse occluded the drains and reopened them when the patient returned to the position described for each group.
  Arms: Trendelenburg

SUMMARY:
Objective: Determine the effect of the postoperative trendelenburg position on the recurrence of chronic subdural hematoma (CSH) in patients undergoing surgery.

Materials and Methods: An open-label, randomized, controlled clinical trial was conducted in three hospitals in Medellín. Patients with CSH were enrolled and assigned to the trendelenburg position (30° leg elevation and 10° head tilt) or a flat bed for 24 hours postoperatively. CSH recurrence was measured at 3 months, along with functional outcome (modified Rankin scale), adverse events, and comfort (Likert scale).

DETAILED DESCRIPTION:
Objective: Determine the effect of the postoperative trendelenburg position on the recurrence of chronic subdural hematoma (CSH) in patients undergoing surgery.

Materials and Methods: An open-label, randomized, controlled clinical trial was conducted in three hospitals in Medellín. Patients with CSH were enrolled and assigned to the trendelenburg position (30° leg elevation and 10° head tilt) or a flat bed for 24 hours postoperatively. CSH recurrence was measured at 3 months, along with functional outcome (modified Rankin scale), adverse events, and comfort (Likert scale).

ELIGIBILITY:
Inclusion Criteria:

* The study included patients aged 18 years or older who required surgical management of symptomatic CSH confirmed by CT scan and whose informed consent was given by the patient or responsible family member to participate in the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Conditions in which the trendelenburg position might not be safe, such as intracranial hypertension without a drain to allow evacuation of the hematoma, cardiovascular instability (severe heart failure, unstable angina, cardiogenic pulmonary edema), acute respiratory distress syndrome without a secure airway, glaucoma, spinal cord trauma not stabilized with surgery, peripheral vascular disease,
* History of ipsilateral chronic subdural hematoma drainage, intracranial hypotension syndrome, ventriculoperitoneal shunting
* Simultaneous participation in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 3 months
  Proportion of patients who experienced recurrence of chronic subdural hematoma at 3 months of follow-up and required repeat surgery

SECONDARY OUTCOMES:
proportion of patients with favorable functional outcome at 3 months, as measured by the modified Rankin Scale. | 3 months
  Secondary outcomes were the proportion of patients with favorable functional outcome at three months, as measured by the modified Rankin Scale (mRS). The validated scale has seven categories: no symptoms (0), no clinically significant disability despite symptoms (1), mild disability (2), moderate disability (3), moderately severe disability (4), severe disability (5), and death (6); in this trial, a score of 0 to 2 was considered a favorable outcome, as it is associated with functional independence.

CONTACTS AND LOCATIONS:
Locations (3):
- Colombia (3):
  - Clinica CES, Medellín, Antioquia
  - Hospital San Vicente Fundación, Medellín, Antioquia
  - Instituto Neurologico de Colombia, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Undecided
It's not clear to me

REFERENCES:
- [Background] Hamou H, Alzaiyani M, Pjontek R, Kremer B, Albanna W, Ridwan H, Clusmann H, Hoellig A, Veldeman M. Risk factors of recurrence in chronic subdural hematoma and a proposed extended classification of internal architecture as a predictor of recurrence. Neurosurg Rev. 2022 Aug;45(4):2777-2786. doi: 10.1007/s10143-022-01790-8. Epub 2022 Apr 23. PMID 35461433